CLINICAL TRIAL: NCT03873428
Title: Evaluation of the Unconformity of the Hormonal Status of Metastatic Lesions During a First Relapse of Breast Cancer Initially Expressing Estrogen Receptors: a Pilot Study on the Interest of Positron Emission Tomography (PET) With 16α- [18F] -Fluoro-17β-estradiol (FES).
Brief Title: Evaluation of the Unconformity of the Hormonal Status of Metastatic Lesions During a First Relapse of Breast Cancer Initially Expressing Estrogen Receptors: a Pilot Study on the Interest of PET With FES
Acronym: EstroTEPCompar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EstroTEP COMPARE
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: FES TEP in Detection of Estrogen Receptors
Keywords: breast cancer; first metastatic relapse; PET
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES PET (Other): 1 ) inclusion; 2 ) FGD PET / FES PET; 3) Hormone therapy
  Interventions: Other: FES PET

INTERVENTIONS:
Other: FES PET — FES injection

SUMMARY:
Breast cancer is a major public health issue despite therapeutic advances, it is the first cause of death cancer of women in Europe.

Several treatments may be proposed depending on the general condition of the patient, the characteristics of the initial tumor and the stage of the disease. The different treatments in metastatic relapse of hormone receptor-positive breast cancer are systemic treatments, such as hormone therapy, chemotherapy, targeted therapies, and possible supportive care, but also in some cases local treatments such as surgery and radiotherapy.

Comparative analysis of primary mammary tumors and their metastases has demonstrated the essential role of tumor heterogeneity, both in time and space, in the progression of the disease and the occurrence of resistance to treatments. Taking into account this intratumoral heterogeneity represents a major axis of improvement in the management of patients with breast cancer.

The use of innovative radiotracers such as 16α- [18F] -fluoro-17β-estradiol (FES) may allow in the future to better evaluate this tumor heterogeneity in patients with metastatic breast cancer through non-metastatic characterization. invasive different lesions. It will be possible to propose to each patient a more personalized care with possibly the administration, in addition to the systemic treatment, of a local treatment adapted to the characteristics of some secondary lesions likely to respond less well to the systemic treatment.

In this pilot study, the investigators would like to estimate the number of patients and the number of metastatic sites affected by tumor heterogeneity of estrogen receptor expression, which could benefit from specific management.

This study will concern a population of patients with first metastatic recurrence of hormone receptor-positive breast cancer initially, with at least one metastasis, who are candidates for treatment with hormone therapy.

DETAILED DESCRIPTION:
The main objective of this pilot study is to determine the unconformity rates for estrogen receptor expression in different metastatic lesions in patients with first metastatic recurrence of breast cancer initially expressing estrogen receptors.

Secondary objectives are:

1. To study the influence of the FES PET could have for possible modifications of therapeutic management in these patients.
2. Determine the rate of patients with additional positive FES lesions but without positive FDG lesions.
3. Evaluate the response to chemotherapy at 3 months after using FDG-PET in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG score (Eastern Cooperative Oncology Group) ≤ 2.
2. Stage IV breast cancer (AJCC TNM).
3. Primitive tumor expressing RO (> 10%).
4. Patient candidate for hormone therapy treatment targeting estrogen receptors as a first-line treatment in a context of first metastatic recurrence.
5. No overexpression of HER2 in the tumor.
6. Lack of previous treatment for metastatic disease
7. Metastatic status confirmed by 18F-FDG PET / CT performed in the month prior to inclusion
8. Life expectancy estimated at more than 3 months.
9. Patient able to understand and give informed informed consent for participation in the study.
10. Patient affiliated with the social security scheme or equivalent.

Exclusion Criteria:

1. Triple negative breast cancer
2. Overexpression HER2 +++
3. Metastatic involvement exclusively in the liver
4. Unable to lie down or maintain the position during the PET / CT scan
5. Uncontrolled intercurrent pathology that is life-threatening in the short term
6. Uncontrolled diabetes
7. History of an allergic reaction attributed to a chemical or biological compound related to FDG or FES
8. Psychiatric impairment or social conditions that would limit patient availability and compliance at different stages of the study.
9. Pregnant woman (mandatory pregnancy test at baseline) or who is breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-10-18 (Estimated); Study Completion 2025-10-18 (Estimated)

PRIMARY OUTCOMES:
Estrogen Receptor Gene Expression | at the inclusion
  number of FDG+ / FES- lesions compared to the number of FDG+ / FES+ lesions

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Georges-François Leclerc, Dijon, Bourgogne-Franche-Comté
  - CGFL, Dijon